CLINICAL TRIAL: NCT04781816
Title: Randomized, Double-blind, Placebo Controlled, Proof of Concept Study Assessing the Efficacy and Safety of the RIPK1-inhibitor SAR443122 in Patients With Moderate to Severe Subacute or Discoid/Chronic Cutaneous Lupus Erythematosus
Brief Title: Proof of Concept Study of SAR443122 in Patients With Cutaneous Lupus Erythematosus
Acronym: CLEan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT16404; U1111-1246-6784 (Registry Identifier: ICTRP); 2020-004703-14 (EudraCT Number)
Record Dates: First submitted 2021-02-28; First posted 2021-03-04 (Actual); Results first posted 2024-06-24 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Cutaneous Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SAR443122 (Experimental): SAR443122 for 12 weeks
  Interventions: Drug: SAR443122
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR443122 — Pharmaceutical form: Capsule Route of administration: Oral
  Arms: SAR443122
Drug: Placebo — Pharmaceutical form: Capsule Route of administration: Oral
  Arms: Placebo

SUMMARY:
Primary Objective:

* Assess the efficacy of SAR443122 in cutaneous lupus erythematosus (CLE)

Secondary Objectives:

* Assess the effect of SAR443122 on the physician's global assessment of disease activity (PhysGA - disease activity)
* Assess the effect of SAR443122 on CLE induced itch and overall pain
* Assess the effect of SAR443122 on the proportion of disease activity responders compared to placebo
* Assess the effect of SAR443122 on the CLASI components score
* Assess the effect of SAR443122 on the Investigator's global assessment for CLE (IGA-CLE)
* Assess oral cavities for patients with oral lesions
* Assess the disease specific quality of life (QoL)
* Assess the safety and tolerability of SAR443122 in patients with CLE
* Assess the pharmacokinetics (PK) exposure of SAR443122 in patients with CLE

DETAILED DESCRIPTION:
Total study duration per participant was up 20 weeks including:

* A screening period of up to 4 weeks
* A treatment period of 12 weeks
* A post treatment follow-up period of 4 weeks

ELIGIBILITY:
Inclusion criteria :

* Participants with cutaneous lupus erythematosus either in the form of discoid/chronic cutaneous lupus erythematosus or subacute cutaneous lupus erythematosus for at least 3 months before Screening.
* Participants with histologically confirmed and documented diagnosis within one year prior to Screening or during Screening period prior to randomization.
* Active cutaneous lupus erythematosus skin lesions and a Cutaneous Erythematosus.
* Disease Area and Severity Index activity (CLASI-A) ≥10 both at Screening and Baseline.
* Participant who was candidate for systemic treatment per Investigator's judgement.

Exclusion criteria:

* Systemic lupus erythematosus according to the 2012 SLICC criteria with major organ involvement.
* Suspected or proven drug induced lupus erythematosus, including patients with positive antihistone autoantibody tests.
* Autoimmune disease(s) other than systemic lupus erythematosus.
* Active skin diseases that may interfere with the study or study assessments.
* Exclusion related to tuberculosis, non-tuberculous mycobacterial infections, HIV, HBV, HCV, Herpes zoster, COVID-19 and other recurrent or recent serious infections.
* Prolonged QTcF ≥ 450 ms (by Fridericia formula) or clinically significant findings on electrocardiogram (ECG).
* Cannot avoid excessive UV exposure 4 weeks prior to baseline and during the study. Routine sun exposure through work are permitted but requires the use of sun block to sun exposed areas for at least 4 weeks prior to baseline and during the study.
* Concomitant treatment with topical immunosuppressants beyond a stable regimen of low to medium potency topical corticosteroids and/or topical calcineurin inhibitors during the study and two weeks before baseline visit.
* Initiation and/or changes in dosage of chloroquine/hydroxychloroquine within 12 weeks prior to Screening visit (or during Screening period) and/or the dose exceeding 2.3 mg/kg/day for chloroquine or 400 mg/day for hydroxychloroquine.
* Systemic treatments for cutaneous or systemic lupus erythematosus or immunosuppressive therapy for autoimmune disease other than the study medication.
* Systemic corticosteroids treatment <4 weeks before baseline visit.
* Live vaccine(s) within 1 month prior to Screening, or plans to receive such vaccines during the study.
* Laboratory abnormalities at the Screening visit.

The above information was not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (50):
- United States (4):
  - GNP Research Site Number : 8400008, Cooper City, Florida
  - DJL Clinical Research, PLLC Site Number : 8400003, Charlotte, North Carolina
  - ClinOhio Research Services Site Number : 8400007, Columbus, Ohio
  - Prolato Clinical Research Center Site Number : 8400010, Houston, Texas
- Argentina (5):
  - Investigational Site Number : 0320002, CABA, Buenos Aires
  - Investigational Site Number : 0320003, CABA, Buenos Aires
  - Investigational Site Number : 0320001, CABA, Buenos Aires
  - Investigational Site Number : 0320004, Rosario, Santa Fe Province
  - Investigational Site Number : 0320005, Mendoza
- Australia (2):
  - Investigational Site Number : 0360001, Camberwell, Victoria
  - Investigational Site Number : 0360002, East Melbourne, Victoria
- Canada (3):
  - Investigational Site Number : 1240001, London, Ontario
  - Investigational Site Number : 1240005, Toronto, Ontario
  - Investigational Site Number : 1240002, Sherbrooke, Quebec
- Chile (6):
  - Investigational Site Number : 1520009, Valdivia, Los Ríos Region
  - Investigational Site Number : 1520006, Osorno, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520007, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
- Czechia (4):
  - Investigational Site Number : 2030002, Brno
  - Investigational Site Number : 2030004, Náchod
  - Investigational Site Number : 2030006, Pardubice
  - Investigational Site Number : 2030005, Prague
- Hungary (2):
  - Investigational Site Number : 3480001, Budapest
  - Investigational Site Number : 3480002, Szeged
- India (3):
  - Investigational Site Number : 3560002, Chandigarh
  - Investigational Site Number : 3560003, Nagpur
  - Investigational Site Number : 3560004, Nashik
- Italy (2):
  - Investigational Site Number : 3800001, Genova
  - Investigational Site Number : 3800002, Milan
- Mexico (4):
  - Investigational Site Number : 4840003, Benito Juárez
  - Investigational Site Number : 4840004, Chihuahua City
  - Investigational Site Number : 4840001, Monterrey, Nuevo León
  - Investigational Site Number : 4840002, Veracruz
- Poland (3):
  - Investigational Site Number : 6160006, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6160004, Lublin, Lublin Voivodeship
  - Investigational Site Number : 6160007, Katowice, Silesian Voivodeship
- Russia (5):
  - Investigational Site Number : 6430004, Krasnodar
  - Investigational Site Number : 6430005, Moscow
  - Investigational Site Number : 6430002, Moscow
  - Investigational Site Number : 6430001, Saint Petersburg
  - Investigational Site Number : 6430003, Stavropol
- Spain (4):
  - Investigational Site Number : 7240002, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240007, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240001, L'Hospitalet de Llobregat, Barcelona [Barcelona]
  - Investigational Site Number : 7240004, Madrid, Madrid, Comunidad de
- Ukraine (2):
  - Investigational Site Number : 8040001, Ivano-Frankivsk
  - Investigational Site Number : 8040002, Kyiv
- Investigational Site Number : 8260003, London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT16404 Cutaneous Lupus Erythematosus website — https://www.sanofistudies.com/1QVB/
- See also: ACT16404 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25191&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 50 centers in 15 countries. A total of 132 participants were screened from 01 April 2021 to 01 March 2023, of which 54 were screen failures. Screen failures were mainly due to not meeting the eligibility criteria.
Pre-assignment Details: A total of 78 participants were randomized in a ratio of 1:1 to either SAR443122 or placebo arm. The randomization was stratified by subtype of cutaneous lupus erythematosus (CLE) (discoid lupus erythematosus [DLE] or subacute cutaneous lupus erythematosus [SCLE]), baseline use of hydroxychloroquine/chloroquine (HCQ/CQ) and by region.
Groups:
- Placebo: Participants received placebo matched to SAR443122 orally twice a day (BID) for 12 weeks.
- SAR443122: Participants received SAR443122 300 mg orally BID for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | SAR443122
Started | 40 | 38
Completed | 38 | 35
Not Completed | 2 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Not Related to Coronavirus Disease 2019 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants exposed to the investigational medicinal product (IMP) (regardless of the amount of treatment administered).
Groups:
- Placebo: Participants received placebo matched to SAR443122 orally BID for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | SAR443122 | Total
Number analyzed (Participants) | 40 | 38 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (9.8) | 45.6 (10.7) | 45.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 33 | 62
  Male | 11 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 7
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 31 | 30 | 61
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Cutaneous Erythematosus Disease Area and Severity Index - Activity (CLASI-A) Sub-Score at Week 12
Description: The CLASI is a clinician rated scale designed to assess the disease activity and damage in CLE in adults. It is composed of 56 items covering 2 dimensions: the disease activity (CLASI-A) and the disease damage (CLASI-D). CLASI-A disease activity covers the domains: erythema, scale/hypertrophy, recent hair loss/alopecia, and mucous membrane lesions. CLASI-A sub-score ranges for 0 to 70, where 0-9 indicates mild disease, 10-20 indicates moderate disease, and 21-70 indicates severe disease. Higher score indicates a more severe skin disease. Baseline was defined as the Day 1 assessment value.
Time Frame: Baseline (Day 1) and Week 12
Population: Efficacy population included all randomized participants exposed to the IMP, with available Baseline assessment of the CLASI-A who actually received at least 1 complete dose of IMP and with at least 1 post IMP administration measurement. Only participants with data collected at Week 12 are reported.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | SAR443122
Number analyzed (Participants) | 35 | 35
percent change | -37.05 (5.31) | -42.76 (5.42)
Statistical Analysis 1: Comparison: Placebo vs SAR443122; Analysis was performed using mixed model with repeated measurements (MMRM) including fixed effects for baseline CLASI-A, post-baseline visit, geographical region, disease subtype, baseline use of CQ/HCQ, intervention group, visit-by- intervention group interaction, and visit-by-baseline-CLASI-A interaction; Test type: Superiority; Least Square Mean Difference = -5.70, 90% CI 2-sided [-18.26 to 6.85], Standard Error of Mean 7.53

2. Secondary Outcome: Percentage of Participants With Physician's Global Assessment of Disease Activity (PhysGA- Disease Activity) of 0 or 1 (Disease Free or Almost Disease Free) at Week 12
Description: The PhysGA- disease activity is a 5 point-Lickert scale instrument designed to assess physician-reported disease activity. The investigators were asked the following question "How active would you say your patient's cutaneous lupus erythematosus is currently?" The total score on scale ranges from 0 (not active at all) to 4 (extremely active). Higher score indicates a more severe skin disease.
Time Frame: Week 12
Population: Efficacy population included all randomized participants exposed to the IMP, with available Baseline assessment of the CLASI-A who actually received at least 1 complete dose of IMP and with at least 1 post IMP administration measurement.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAR443122
Number analyzed (Participants) | 40 | 38
percentage of participants | 32.5 | 44.74

3. Secondary Outcome: Change From Baseline in Participants Reported Daily Worst Itch Using Peak Pruritus Numerical Rating Scale (Itch-NRS) at Week 12
Description: The Peak Pruritus NRS (itch-NRS) is a single item patient reported outcomes (PRO) tool that participants used to report the intensity of their pruritus (itch) during a daily recall period. Participants were asked to rate their worst itch on a 0 (no itch) to 10 (worst itch imaginable) NRS by answering the following question: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". The total score on scale ranges from 0 (no itch) to 10 (worst itch imaginable). Higher score indicates a more severe skin disease. Baseline was defined as the average of daily non-missing scores obtained during the week prior to Day 1.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAR443122
Number analyzed (Participants) | 40 | 36
score on a scale | -0.62 (0.37) | -2.16 (0.39)

4. Secondary Outcome: Change From Baseline in Participants Reported Daily Worst Pain Using Peak Pain Numerical Rating Scale (Pain-NRS) at Week 12
Description: The Peak Pain NRS (Pain-NRS) is a single item PRO tool that participants used to report the intensity of their CLE-related pain (skin, oral, genital) during a daily recall period. Participants were asked to rate their worst pain on a 0 (no pain) to 10 (worst pain imaginable) NRS by answering the following question: "On a scale of 0 to 10, with 0 being 'no pain' and 10 being the 'worst pain imaginable', how would you rate your pain at the worst moment due to your lupus during the previous 24 hours?". The total score on scale ranges from 0 (no pain) to 10 (worst pain imaginable). Higher score indicates a more severe skin disease. Baseline was defined as the average of daily non-missing scores obtained during the week prior to Day 1.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAR443122
Number analyzed (Participants) | 40 | 36
score on a scale | -0.93 (0.32) | -1.72 (0.34)

5. Secondary Outcome: Percentage of CLASI-A50 and CLASI-A75 Responders at Week 12
Description: The CLASI is a clinician rated scale designed to assess the disease activity and damage in CLE in adults. It is composed of 56 items covering 2 dimensions: the disease activity (CLASI-A) and the disease damage (CLASI-D). CLASI-A disease activity covers the domains: erythema, scale/hypertrophy, recent hair loss/alopecia, and mucous membrane lesions. CLASI-A sub-score ranges for 0 to 70, where 0-9 indicates mild disease, 10-20 indicates moderate disease, and 21-70 indicates severe disease. Higher score indicates a more severe skin disease. The CLASI-A50/75 responder was defined as a participant who achieved a decrease by at least 50%/75% of CLASI-A sub-score from baseline.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of responders
Arm/Group | Placebo | SAR443122
Number analyzed (Participants) | 40 | 38
percentage of responders
  CLASI-A50 | 45 | 44.74
  CLASI-A75 | 10 | 23.68

6. Secondary Outcome: Change From Baseline in CLASI Components' Score Over Time
Description: The CLASI is a clinician rated scale designed to assess the disease activity and damage in CLE in adults. It is composed of 56 items covering two dimensions: the disease activity (CLASI-A) and the disease damage (CLASI-D). CLASI-A disease activity covers the domains: erythema, scale/hypertrophy, recent hair loss/alopecia, and mucous membrane lesions. CLASI-A sub-score ranges 0 to 70, where 0-9 indicates mild disease, 10-20 indicates moderate disease, and 21-70 indicates severe disease. CLASI-D disease damage covers the domains: dyspigmentation, scarring/atrophy/panniculitis, and clinically judged scarring of the scalp (including scarring alopecia). Scale ranges 0 (absence of disease damage) to 56 (severe disease damage) using the parameters of dyspigmentation and scarring. For CLASI-A and CLASI-D, higher score indicates a more severe skin disease. Change from baseline in CLASI components' score are reported. Baseline was defined as the Day 1 assessment value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, and 16
Population: Efficacy population included all randomized participants exposed to the IMP, with available Baseline assessment of the CLASI-A who actually received at least 1 complete dose of IMP and with at least 1 post IMP administration measurement. Only participants with data collected at Weeks 4, 8, 12, and 16 for each specified category are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | SAR443122
Number analyzed (Participants) | 40 | 38
score on a scale
  Erythema: Weeks 4: number analyzed (Participants) | 40 | 37
  Erythema: Weeks 4 | -2.33 (3.24) | -2.14 (3.02)
  Erythema: Weeks 8: number analyzed (Participants) | 38 | 36
  Erythema: Weeks 8 | -3.37 (4.48) | -3.42 (3.80)
  Erythema: Weeks 12: number analyzed (Participants) | 35 | 35
  Erythema: Weeks 12 | -4.97 (4.89) | -4.17 (4.15)
  Erythema: Weeks 16: number analyzed (Participants) | 34 | 33
  Erythema: Weeks 16 | -5.09 (4.00) | -4.18 (4.38)
  Scale/Hypertrophy: Week 4: number analyzed (Participants) | 40 | 37
  Scale/Hypertrophy: Week 4 | -0.83 (1.32) | -1.86 (2.47)
  Scale/Hypertrophy: Week 8: number analyzed (Participants) | 38 | 36
  Scale/Hypertrophy: Week 8 | -1.34 (2.34) | -2.72 (3.19)
  Scale/Hypertrophy: Week 12: number analyzed (Participants) | 35 | 35
  Scale/Hypertrophy: Week 12 | -2.03 (2.99) | -3.17 (3.34)
  Scale/Hypertrophy: Week 16: number analyzed (Participants) | 34 | 33
  Scale/Hypertrophy: Week 16 | -2.12 (2.58) | -3.30 (3.54)
  Scarring/Atrophy/Panniculitis: Week 4: number analyzed (Participants) | 40 | 37
  Scarring/Atrophy/Panniculitis: Week 4 | -0.13 (0.88) | -0.16 (0.83)
  Scarring/Atrophy/Panniculitis: Week 8: number analyzed (Participants) | 38 | 36
  Scarring/Atrophy/Panniculitis: Week 8 | -0.08 (1.08) | -0.25 (0.87)
  Scarring/Atrophy/Panniculitis: Week 12: number analyzed (Participants) | 35 | 35
  Scarring/Atrophy/Panniculitis: Week 12 | -0.06 (1.37) | -0.06 (1.26)
  Scarring/Atrophy/Panniculitis: Week 16: number analyzed (Participants) | 34 | 33
  Scarring/Atrophy/Panniculitis: Week 16 | -0.24 (1.48) | -0.18 (1.26)

7. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment of Cutaneous Lupus Erythematosus (IGA-CLE) Score of 0 or 1 (Clear Or Almost Clear) at Week 12
Description: The IGA-CLE is a clinician reported outcome (ClinRO) that allows for clinicians to assess the overall disease activity of CLE using a 5-point scale: 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate), and 4 (severe). The severity of CLE is determined by descriptions of a combination of 3 plaque characteristics: erythema, scale, elevation. Erythema is the primary characteristic that influenced the rating, with other characteristics considered secondarily. Telangiectatic change is not considered in the rating. The assessment did not require the presence of all 4 characteristics, the severity was averaged over the observed characteristics. The total score on scale ranges from 0 to 4. Higher score indicates a more severe skin disease.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAR443122
Number analyzed (Participants) | 38 | 34
percentage of participants | 15.79 | 26.47

8. Secondary Outcome: Change From Baseline to Week 12 in the Oral Health Impact Profile 14-Item Version (OHIP-14) for Participants With Oral Lesions at Baseline
Description: The OHIP-14 is a PRO questionnaire that is composed of 14 items that assess 7 different dimensions, considering the perception of the individual in relation to the impact of oral conditions in the physical, psychological and social well-being in the last month. Each of the 14 items has a set of possible answers distributed in a Likert scale (0 = never, 1 = hardly ever. 2 = occasionally 3 = fairly often, 4 = very often), which represents the frequency that the individual perceives the impact of oral health on 7 dimensions: functional limitation (2 items), physical pain (2 items), psychological discomfort (2 items), physical disability (2 items), psychological disability (2 items), social disability (2 items) and handicap (2 items). The OHIP-14 scores range from 0 to 56 and are calculated by summing the ordinal values for 14 items. Domain scores range from 0 to 8. Higher OHIP-14 scores indicate worse oral-health-related quality of life. Baseline was defined as Day 1 assessment value.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | SAR443122
Number analyzed (Participants) | 10 | 13
score on a scale | -2.90 (7.68) | -0.15 (4.79)

9. Secondary Outcome: Change From Baseline in SKINDEX-29+3 Total Score at Week 12
Description: Skindex 29+3 is a PRO measure designed to assess the effects of skin disease on participants' health-related quality of life in adults. It contains the following domains: emotions (10 items), symptoms (7 items), functioning (12 items), lupus-specific issues (3 questions), and 1 item about treatment that is not part of the total score. Recall period is during the past week. Each item is rated on a 5-point Likert scale (never, rarely, sometimes, often, all the time). These responses are then transformed to a linear scale ranging from 0 to 100 in 25-point increments, with 100 representing maximal disability. The total score is the average of participants' responses to items in a given domain, ranging from 0 to 100, where higher scores indicate a greater impact on the health-related quality of life. Baseline was defined as the Day 1 assessment value.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAR443122
Number analyzed (Participants) | 40 | 38
score on a scale | -9.09 (2.31) | -11.09 (2.35)

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Treatment-emergent Serious Adverse Events (TESAEs), and Adverse Events of Special Interest (AESIs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAEs were defined as the adverse events that occurred from the time of the first IMP administration up to the end of study visit. Serious adverse events (SAE): Any AE that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. An AESI: an AE (serious or nonserious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor was required.
Time Frame: From first dose of study treatment (Day 1) up to end of study (Week 16)
Population: Safety population included all randomized participants exposed to the IMP (regardless of the amount of treatment administered).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAR443122
Number analyzed (Participants) | 40 | 38
Participants
  Any TEAE | 18 | 22
  Any TESAE | 1 | 0
  Any AESI | 1 | 2

11. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities (PCSA) in Hematology Parameters
Description: PCSA values were defined as abnormal values considered medically important by the Sponsor, according to predefined criteria/thresholds based on literature reviews and defined by the Sponsor. Criteria for PCSA: Hemoglobin (Hb) ≤ 115 grams per liter (g/L) (Male [M]) or ≤ 95 g/L (Female [F]), ≥ 185 g/L (M) or ≥ 165 g/L (F), decrease from baseline ≥ 20 g/L; Platelets <100 x 10^9 per liter (/L) or ≥ 700 x 10^9/L; Erythrocytes ≥ 6 x 10^12/L; Leukocytes < 3 x 10^9/L (Non-Black [NB]); < 2 x 10^9/L (Black[B]); or ≥ 16 x 10^9/L; Neutrophils < 1.5 x 10^9/L (NB); < 1 x 10^9/L (B); Lymphocytes > 4 x 10^9/L; Monocytes > 0.7 x 10^9/L; Basophils > 0.1 x 10^9/L; Eosinophils > 0.5 x 10^9/L or > upper limit of normal range (ULN) (if ULN ≥ 0.5 x 10^9/L).
Time Frame: From first dose of study treatment (Day 1) up to end of study (Week 16)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAR443122
Number analyzed (Participants) | 40 | 38
Participants
  Hb: ≤ 115 g/L (M); ≤ 95 g/L (F) | 0 | 1
  Hb: ≥ 185 g/L (M); ≥ 165 g/L (F) | 0 | 0
  Decrease from baseline ≥ 20 g/L | 0 | 0
  Platelets < 100 x 10^9/L | 0 | 0
  Platelets ≥ 700 x 10^9/L | 0 | 0
  Erythrocytes ≥ 6 x 10^12/L | 0 | 0
  Leukocytes < 3 x 10^9/L (NB); < 2 x 10^9/L (B) | 3 | 0
  Leukocytes ≥ 16 x 10^9/L | 0 | 0
  Neutrophils < 1.5 x 10^9/L (NB); < 1 x 10^9/L (B) | 3 | 0
  Lymphocytes > 4 x 10^9/L | 0 | 0
  Monocytes > 0.7 x 10^9/L | 1 | 3
  Basophils > 0.1 x 10^9/L | 6 | 5
  Eosinophils > 0.5 x 10^9/L or > ULN | 1 | 1

12. Secondary Outcome: Number of Participants With PCSA in Clinical Chemistry
Description: PCSA values were defined as abnormal values considered medically important by the Sponsor, according to predefined criteria/thresholds based on literature reviews and defined by the Sponsor. Criteria for PCSA: Glucose ≤ 3.9 millimoles per liter (mmol/L) and < lower limit of normal range (LLN) or ≥ 11.1 mmol/L (unfasted); ≥ 7 mmol/L (fasted); Creatine Kinase > 3 ULN; Sodium ≤ 129 mmol/L or ≥ 160 mmol/L; Potassium < 3 mmol/L or ≥ 5.5 mmol/L; Creatinine ≥ 150 micromoles per liter (μmol/L) (Adults) or ≥ 30% change from baseline or ≥ 100% change from baseline; Creatinine Clearance ≥ 60 - < 90 milliliters per minute (mL/min) (mild decrease in glomerular filtration rate [GFR]) or ≥ 30 - < 60 mL/min (moderate decrease in GFR) or ≥ 15 - < 30 mL/min (severe decrease in GFR) or < 15 mL/min (end stage renal disease); Alanine Aminotransferase > 3 ULN or > 5 ULN; Aspartate Aminotransferase > 3 ULN or > 5 ULN; Alkaline Phosphatase > 1.5 ULN; Total Bilirubin > 1.5 ULN.
Time Frame: From first dose of study treatment (Day 1) up to end of study (Week 16)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAR443122
Number analyzed (Participants) | 40 | 38
Participants
  Glucose ≤ 3.9 mmol/L and < LLN | 4 | 1
  Glucose ≥11.1 mmol/L(unfasted); ≥7mmol/L(fasted) | 1 | 3
  Creatine Kinase > 3 ULN | 0 | 0
  Sodium ≤ 129 mmol/L | 0 | 0
  Sodium ≥ 160 mmol/L | 0 | 0
  Potassium < 3 mmol/L | 0 | 0
  Potassium ≥ 5.5 mmol/L | 2 | 0
  Creatinine ≥ 150 μmol/L (Adults) | 0 | 0
  Creatinine ≥ 30% change from baseline | 2 | 1
  Creatinine ≥ 100% change from baseline | 0 | 0
  Creatinine Clearance ≥ 60 - < 90 mL/min | 10 | 8
  Creatinine Clearance ≥ 30 - < 60 mL/min | 0 | 0
  Creatinine Clearance ≥ 15 - < 30 mL/min | 0 | 0
  Creatinine Clearance < 15 mL/min | 0 | 0
  Alanine Aminotransferase > 3 ULN | 1 | 2
  Alanine Aminotransferase > 5 ULN | 0 | 0
  Aspartate Aminotransferase > 3 ULN | 1 | 0
  Aspartate Aminotransferase > 5 ULN | 0 | 0
  Alkaline Phosphatase > 1.5 ULN | 5 | 0
  Total Bilirubin > 1.5 ULN | 0 | 0

13. Secondary Outcome: Number of Participants With PCSA in Urinalysis
Description: PCSA values were defined as abnormal values considered medically important by the Sponsor, according to predefined criteria/thresholds based on literature reviews and defined by the Sponsor. Criteria for PCSA: pH ≤ 4.6 or ≥ 8.
Time Frame: From first dose of study treatment (Day 1) up to end of study (Week 16)
Population: Safety population included all randomized participants exposed to the IMP (regardless of the amount of treatment administered). Only participants with data collected for each specified category at Week 16 are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAR443122
Number analyzed (Participants) | 40 | 38
Participants
  pH ≤ 4.6: number analyzed (Participants) | 39 | 38
  pH ≤ 4.6 | 0 | 0
  pH ≥ 8: number analyzed (Participants) | 39 | 38
  pH ≥ 8 | 0 | 0

14. Secondary Outcome: Number of Participants With PCSA in Electrocardiogram (ECG)
Description: PCSA values were defined as abnormal values considered medically important by the Sponsor, according to predefined criteria/thresholds based on literature reviews and defined by the Sponsor. Criteria for PCSA: Heart Rate (HR) < 50 beats/min (bpm) or < 50 bpm and decrease from baseline ≥ 20 bpm or < 40 bpm or > 90 bpm; PR Interval > 200 milliseconds (msec) or > 200 msec and increase from baseline ≥ 25% or > 220 msec; QRS Interval > 110 msec or 110 msec and increase from baseline ≥ 25% or > 120 msec; QT Interval > 500 msec; corrected QT (QTc) Interval > 450 msec or > 480 msec or increase from baseline [30-60] msec or increase from baseline > 60 msec.
Time Frame: From first dose of study treatment (Day 1) up to end of study (Week 16)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAR443122
Number analyzed (Participants) | 40 | 38
Participants
  HR < 50 bpm: number analyzed (Participants) | 36 | 36
  HR < 50 bpm | 2 | 1
  HR < 50 bpm and decrease from baseline ≥ 20 bpm: number analyzed (Participants) | 36 | 36
  HR < 50 bpm and decrease from baseline ≥ 20 bpm | 0 | 0
  HR < 40 bpm: number analyzed (Participants) | 36 | 36
  HR < 40 bpm | 0 | 0
  HR > 90 bpm: number analyzed (Participants) | 36 | 36
  HR > 90 bpm | 2 | 1
  PR Interval > 200 msec: number analyzed (Participants) | 36 | 36
  PR Interval > 200 msec | 2 | 0
  PR Interval >200 msec;increase from baseline ≥25%: number analyzed (Participants) | 36 | 36
  PR Interval >200 msec;increase from baseline ≥25% | 0 | 0
  PR Interval > 220 msec: number analyzed (Participants) | 36 | 36
  PR Interval > 220 msec | 0 | 0
  QRS Interval > 110 msec: number analyzed (Participants) | 36 | 36
  QRS Interval > 110 msec | 0 | 2
  QRS Interval >110 msec;increase from baseline≥25%: number analyzed (Participants) | 36 | 36
  QRS Interval >110 msec;increase from baseline≥25% | 0 | 0
  QRS Interval > 120 msec: number analyzed (Participants) | 36 | 36
  QRS Interval > 120 msec | 0 | 0
  QT Interval > 500 msec: number analyzed (Participants) | 36 | 36
  QT Interval > 500 msec | 1 | 0
  QTc Interval > 450 msec: number analyzed (Participants) | 36 | 36
  QTc Interval > 450 msec | 1 | 1
  QTc Interval > 480 msec: number analyzed (Participants) | 36 | 36
  QTc Interval > 480 msec | 0 | 0
  QTc Interval: Increase from baseline [30-60] msec: number analyzed (Participants) | 36 | 36
  QTc Interval: Increase from baseline [30-60] msec | 4 | 0
  QTc Interval: Increase from baseline > 60 msec: number analyzed (Participants) | 36 | 36
  QTc Interval: Increase from baseline > 60 msec | 0 | 0

15. Secondary Outcome: Number of Participants With PCSA in Vital Signs
Description: PCSA values were defined as abnormal values considered medically important by the Sponsor, according to predefined criteria/thresholds based on literature reviews and defined by the Sponsor. Criteria for PCSA: Diastolic Blood Pressure (DBP) ≤ 45 millimeters of mercury (mmHg) and decrease from baseline ≥ 10 mmHg or ≥ 110 mmHg and increase from baseline ≥ 10 mmHg; Pulse Rate (PR) ≤ 50 bpm and decrease from baseline ≥ 20 bpm or ≥ 120 bpm and increase from baseline ≥ 20 bpm; Systolic Blood Pressure (SBP) ≤ 95 mmHg and decrease from baseline ≥ 20 mmHg or ≥ 160 mmHg and increase from baseline ≥ 20 mmHg; Weight ≥ 5% decrease from baseline or ≥ 5% increase from baseline.
Time Frame: From first dose of study treatment (Day 1) up to end of study (Week 16)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAR443122
Number analyzed (Participants) | 40 | 38
Participants
  DBP ≤45 mmHg and decrease from baseline ≥10 mmHg | 0 | 1
  DBP ≥110 mmHg and increase from baseline ≥10 mmHg | 0 | 0
  PR ≤ 50 bpm and decrease from baseline ≥ 20 bpm | 0 | 0
  PR ≥ 120 bpm and increase from baseline ≥ 20 bpm | 0 | 0
  SBP ≤95 mmHg; decrease from baseline ≥20 mmHg | 0 | 1
  SBP ≥160 mmHg; increase from baseline ≥20 mmHg | 0 | 0
  Weight ≥ 5% decrease from baseline: number analyzed (Participants) | 38 | 38
  Weight ≥ 5% decrease from baseline | 3 | 5
  Weight ≥ 5% increase from baseline: number analyzed (Participants) | 38 | 38
  Weight ≥ 5% increase from baseline | 1 | 2

16. Secondary Outcome: Maximum Plasma Concentration (Cmax) of SAR443122
Description: Blood samples were collected at the specified timepoints. Cmax was assessed by a Bayesian analysis using the population PK model.
Time Frame: 2-5 hours post first morning dose on Days 1, 57, and 85; 1 hour before morning dose on Days 57 and 85; 7-10 hours after morning dose on Day 57
Population: PK population included all randomized and treated participants for whom the PK data are considered interpretable. Participants with data collected at Day 1, 57, and 85 are reported.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SAR443122
Number analyzed (Participants) | 36
ng/mL
  Day 1 | 3334 (1365)
  Day 57: number analyzed (Participants) | 33
  Day 57 | 4875 (1541)
  Day 85: number analyzed (Participants) | 31
  Day 85 | 4896 (2013)

17. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of SAR443122
Description: Blood samples were collected at the specified timepoints. tmax was assessed by a Bayesian analysis using the population PK model.
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Median (Full Range); unit: hours
Arm/Group | SAR443122
Number analyzed (Participants) | 36
hours
  Day 1 | 2.80 [NA to 4.90] — NA signifies that some tmax values were not calculable for participants with a low compliance, because all concentrations were below the lower limit of quantification.
  Day 57: number analyzed (Participants) | 33
  Day 57 | 2.60 [NA to 4.35] — NA signifies that some tmax values were not calculable for participants with a low compliance, because all concentrations were below the lower limit of quantification.
  Day 85: number analyzed (Participants) | 31
  Day 85 | 2.55 [NA to 4.30] — NA signifies that some tmax values were not calculable for participants with a low compliance, because all concentrations were below the lower limit of quantification.

18. Secondary Outcome: Area Under the Curve From Time 0 to 12 Hours (AUC0-12) of SAR443122
Description: Blood samples were collected at the specified timepoints. AUC0-12 was assessed by a Bayesian analysis using the population PK model.
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | SAR443122
Number analyzed (Participants) | 36
nanogram*hour per milliliter (ng*h/mL)
  Day 1 | 30151 (14926)
  Day 57: number analyzed (Participants) | 33
  Day 57 | 40194 (15831)
  Day 85: number analyzed (Participants) | 31
  Day 85 | 44489 (19232)

19. Secondary Outcome: Terminal Elimination Half-Life (t1/2z) of SAR443122
Description: Blood samples were collected at the specified timepoints. t1/2z was assessed by a Bayesian analysis using the population PK model.
Time Frame: 1 hour before morning dose and 2-5 hours post first morning dose on Day 85
Population: PK population included all randomized and treated participants for whom the PK data are considered interpretable. Participants with data collected at Day 85 are reported.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | SAR443122
Number analyzed (Participants) | 36
hours | 7.62 (2.28)

ADVERSE EVENTS:
Time Frame: From first dose of study treatment (Day 1) up to end of study (Week 16)
Description: Analysis was performed on safety population.
Arm/Group | Placebo | SAR443122
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/38
Other Adverse Events (participants affected / at risk) | 18/40 | 22/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | SAR443122 (N=38)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | SAR443122 (N=38)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coronary Artery Stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Maculopathy (Eye disorders) | 0 (0) | 1 (1)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Influenza Like Illness (General disorders) | 0 (0) | 1 (1)
Peripheral Swelling (General disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0)
Nail Infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3)
Oral Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oral Herpes (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Tinea Pedis (Infections and infestations) | 1 (1) | 0 (0)
Tooth Abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal Mycotic Infection (Infections and infestations) | 1 (1) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Neutrophil Count Decreased (Investigations) | 0 (0) | 1 (1)
Urine Protein/Creatinine Ratio Increased (Investigations) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone Cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tension Headache (Nervous system disorders) | 1 (1) | 1 (1)
Breast Mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cutaneous Lupus Erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT04781816/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT04781816/SAP_001.pdf